CLINICAL TRIAL: NCT00950651
Title: A Comparison of the Analgesic Efficacy and Safety of Once Daily Tramadol HCl / Contramid® Tablets to Twice Daily Tramadol HCl (SR) for the Treatment of Osteoarthritis of the Knee.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Labopharm Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MDT3-001-E1; NCT00950651 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-04-14; First posted 2009-08-03 (Estimated); Results first posted 2009-08-03 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Osteoarthritis, Knee; Pain
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 Tramadol HCl Contramid® Once A Day (Experimental)
  Interventions: Drug: Tramadol HCl Contramid® Once A Day
- 2 Tramadol HCl Twice a day (SR) (Active Comparator)
  Interventions: Drug: Tramadol HCl Twice a day

INTERVENTIONS:
Drug: Tramadol HCl Contramid® Once A Day — The patients orally self-administered the study medication: either 100, 200, 300 or 400 mg Tramadol HCl Contramid® Once A Day. Each patient was titrated to his or her optimum dose (up to a maximum of 400 mg) during the Titration Phase, which lasted between 4 and 12 days. The optimum dose was taken throughout the study.
  Arms: 1 Tramadol HCl Contramid® Once A Day
Drug: Tramadol HCl Twice a day — The patients orally self-administered the study medication: either 200, 300 or 400 mg Tramadol HCl Twice a day. Each patient was titrated to his or her optimum dose (up to a maximum of 400 mg) during the Titration Phase, which lasted between 4 and 12 days. The optimum dose was taken throughout the study.
  Arms: 2 Tramadol HCl Twice a day (SR)

SUMMARY:
A randomised, multi-centre, double-blind, double dummy, two arm parallel design study to compare the efficacy, safety, and clinical benefit of the test and reference product after treatment for 84 days in patients with osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females between the ages of 40 and 75 with a diagnosis of Osteoarthritis (OA) of the knee consistent with the American College of Rheumatology (ACR) Clinical Classification Criteria for Arthritis of the Knee (Altman, R. et al., 1986):

   * Knee pain at study enrolment,
   * Less than 30 minutes of morning stiffness with or without crepitus on active motion.
   * Confirmation either by arthroscopy or radiologist's report (X-rays showing osteophytes, joint space narrowing or subchondral bone sclerosis {eburnation}) within 1 year prior to entry into the study.
2. ESR < 40 mm/h
3. Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Pain Subscales total score equal to or more than 150 mm at baseline.
4. Oral and written language comprehension at a level sufficient to comply with the protocol and complete study-related materials.
5. The Patient signed and dated the (IEC) approved, written, informed consent prior to study participation

Exclusion Criteria:

1. Known rheumatoid arthritis or any other rheumatoid disease.
2. Secondary arthritis i.e. any of the following: septic arthritis; inflammatory joint disease; gout; pseudogout; Paget's disease; joint fracture; acromegaly; fibromyalgia; Wilson's disease; Ochronosis; Haemochromatosis; Osteochondromatosis; heritable arthritic disorders; or collagen gene mutations.
3. Obesity Class II [body mass index (BMI) equal to or more than 35 kg/m2] (NIH, 2000)
4. Major illness that required hospitalisation during the 3 months before commencement of the screening period.
5. Unwillingness to cease taking medication other than the study medication for arthritic pain, any other concomitant pain, or OA medications.
6. Patients who had previously failed tramadol HCl therapy or those who discontinued tramadol HCl due to AEs.
7. Patients who within the 3 weeks prior to study entry took the following medications: monoamine oxidase inhibitors; tricyclic antidepressants and other tricyclic compounds (e.g. cyclobenzaprine, promethazine); neuroleptics; selective serotonin reuptake inhibitors; or other drugs which reduce seizure threshold.
8. Patients who took another investigational agent within the 30 days prior to study entry.
9. Patients with a history of seizure disorder other than Infantile Febrile Seizures.
10. Patients who were opioid dependent.
11. Patients with bowel disease causing malabsorption.
12. Patients who were pregnant or lactating or patients of child-bearing potential who were unwilling to utilise a medically approved method of contraception during participation in this clinical trial.
13. Patients with significant liver disease, defined as active hepatitis or elevated liver enzymes >3 times the upper boundary of the normal range.
14. Patients with significant renal disease, defined as creatinine clearance <30 mL/min as estimated by the method of Levey et al., 1999.
15. Current substance abuse or dependence, other than nicotine.
16. Allergy or adverse reaction to tramadol or any structurally similar drugs e.g. opiates.
17. Any other condition that, in the opinion of the investigators, adversely affected the patient's ability to complete the study or its measures.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 431 (Actual)
Dates: Start 2002-03; Primary Completion 2002-11 (Actual); Study Completion 2002-11 (Actual)

REFERENCES:
- [Result] Mongin G, Yakusevich V, Kope A, Shostak N, Pikhlak E, Popdan L, Simon J, Navarro C, Fortier L, Robertson S, Bouchard S. Efficacy and Safety Assessment of a Novel Once-Daily Tablet Formulation of Tramadol : A Randomised, Controlled Study versus Twice-Daily Tramadol in Patients with Osteoarthritis of the Knee. Clin Drug Investig. 2004;24(9):545-58. doi: 10.2165/00044011-200424090-00005. PMID 17523716

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol HCl Contramid® Once A Day: The available doses for Tramadol HCl Contramid Once A Day (OAD) were 100 mg, 200 mg, 300 mg or 400 mg daily. Each patient was titrated to his/her optimum dose (based on efficacy and tolerability) and maintained that dose until the end of the study.
- Tramadol HCl Twice a Day (SR): The available doses for Tramadol HCl Twice a day (SR) were 200 mg, 300 mg or 400 mg daily. Each patient was titrated to his/her optimum dose (based on efficacy and tolerability) and maintained that dose until the end of the study.
Period: Overall Study
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Started | 215 | 216 (216 patients randomized but one never took study medication)
Completed | 184 | 181
Not Completed | 31 | 35
Not completed — Adverse Event | 17 | 20
Not completed — Death | 1 | 0
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 3 | 4
Not completed — Withdrawal by Subject | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR) | Total
Number analyzed (Participants) | 215 | 215 | 430
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 121 | 137 | 258
  >=65 years | 94 | 78 | 172
Age Continuous [Mean (Standard Deviation); unit: years] | 61.9 (8.8) | 59.9 (9.1) | 60.9 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 176 | 357
  Male | 34 | 39 | 73

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change From Baseline in WOMAC Pain Subscale Score at Week 12
Description: The WOMAC is a statistically validated, 24-item questionnaire assessing current OA symptoms and functional limitations. The Pain subscale score consists of 5 items each rated on a 100mm VAS scale (0mm=no pain to 100mm=extreme pain). In case of premature discontinuation, the last assessment was used to calculate the percentage of change.
Time Frame: Baseline to week 12
Population: Per protocol population: patients who completed study, had no major protocol deviations before/during trial and had primary efficacy variable rating at end of study. Early drop-outs due to AEs / lack of efficacy were included if they took study drug for >2weeks in maintenance phase and had efficacy assessments within 2 days after end of study drug.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 58.3 (29.9) | 58.7 (27.0)

2. Secondary Outcome: Arthritis Pain at the End of Dosing Interval (24-hour Efficacy)
Description: Each day before morning dose, patients assessed arthritis pain in worst knee in a diary using a 5-point rating scale ranging from none to severe. A median score was estimated for each patient each week and re-categorized into different degrees of pain (rounding off to the closest integer). Results are of 12th week (day 78-84).
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  None | 20 | 19
  Barely noticeable | 42 | 33
  Mild | 35 | 40
  Moderate | 35 | 32
  Severe | 2 | 5

3. Secondary Outcome: Percentage of Change From Baseline in WOMAC Stiffness Subscale Score at Week 12
Description: The WOMAC is a statistically validated, 24-item questionnaire assessing current OA symptoms and functional limitations. Stiffness subscale score consists of 2 items each rated on 100mm VAS scale (0mm=no stiffness to 100mm=extreme stiffness). In case of premature discontinuation, the last assessment was used to calculate the percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 49.1 (60.8) | 49.5 (37.9)

4. Secondary Outcome: Percentage of Change From Baseline in WOMAC Physical Function Subscale Score at Week 12
Description: The WOMAC is a statistically validated, 24-item questionnaire assessing current OA symptoms and functional limitations. Physical Function subscale score consists of 17 items rated on a 100mm VAS scale (0mm=no difficulty to 100mm=extreme difficulty). In case of premature discontinuation, the last assessment was used to calculate percentage of change
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 50.8 (32.5) | 49.8 (29.7)

5. Secondary Outcome: Percentage of Change From Baseline in WOMAC Total Score at Week 12
Description: The WOMAC is a statistically validated, 24-item questionnaire assessing current OA symptoms and functional limitations. Each item is rated on a 100mm VAS scale (0mm=no pain/stiffness/difficulty to 100mm=extreme no pain/stiffness/difficulty). In case of premature discontinuation, the last assessment was used to calculate percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 52.9 (30.9) | 52.0 (28.5)

6. Secondary Outcome: Percentage of Change From Baseline in Current Pain at Week 12
Description: Pain Visual Analogue Scales: Current Pain. Patients indicated their current pain using a 100mm VAS scale ranging from 0=no pain to 100=extreme pain. The percentage of change in current pain was calculated from baseline to week 12. In case of premature discontinuation, the last assessment was used to calculate percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 35.1 (23.8) | 34.6 (23.5)

7. Secondary Outcome: Percentage of Change From Baseline in Least Pain Within Last 24 Hours at Week 12
Description: Patients indicated their Least Pain Within Last 24 Hours using a 100mm VAS scale ranging from 0=no pain to 100=extreme pain. The percentage of change was calculated from baseline to week 12. In case of premature discontinuation, the last assessment was used to calculate percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 21.6 (21.3) | 23.5 (21.2)

8. Secondary Outcome: Percentage of Change From Baseline in Worst Pain Within Last 24 Hours at Week 12
Description: Patients indicated their Worst Pain Within Last 24 Hours using a 100mm VAS scale ranging from 0=no pain to 100=extreme pain. The percentage of change was calculated from baseline to week 12. In case of premature discontinuation, the last assessment was used to calculate percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 38.6 (27.9) | 39.2 (26.3)

9. Secondary Outcome: Percentage of Change From Baseline in Average Pain Within Last 24 Hours at Week 12
Description: Patients indicated their Average Pain Within Last 24 Hours using a 100mm VAS scale ranging from 0=no pain to 100=extreme pain. The percentage of change was calculated from baseline to week 12. In case of premature discontinuation, the last assessment was used to calculate percentage of change.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 30.1 (22.0) | 30.7 (19.7)

10. Secondary Outcome: Percentage of Change From Baseline in Walking Time for 15 Meters at Week 12
Description: The walking test is a measure of how many seconds it takes the patient to walk a distance of 15 meters. The change from baseline to week 12 was calculated.
Time Frame: Baseline to week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
percentage of change | 5.639 (6.231) | 4.738 (5.495)

11. Secondary Outcome: Patient Global Rating of Pain Relief at Week 12
Description: The Patient Global Rating of Pain is a Likert-scale that answers the question: "How do you rate overall pain relief with the drug?" with 4 possible answers that were dichotomized: "very effective", "effective", and "somewhat effective" were summarized to "effective"; "not effective" remained unchanged.
Time Frame: 12 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Effective | 160 | 151
  Not effective | 1 | 2

12. Secondary Outcome: Patient Global Assessment: Side Effects Interfering With Day to Day Activities at Week 12
Description: Patients were asked: "How have any side effects you may have felt from the drug interfered with day-to-day activities?" with 4 possible answers: "Significantly", "Somewhat", "Minimally", "Not at all".
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Significantly | 7 | 2
  Somewhat | 15 | 18
  Minimally | 39 | 34
  Not at all | 100 | 99

13. Secondary Outcome: Patient Global Assessment: Current Pain Relief Versus Pain Relief During Previous Tramadol Treatment at Week 12
Description: Patients who have previously taken tramadol HCl were asked to compare how they compare the current pain relief to the pain relief felt when previously taking tramadol, using a 4-point Likert-scale: "Worse than before", "Same as before", "Somewhat better now", or "Much better now".
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Worse than before | 0 | 0
  Same as before | 4 | 2
  Somewhat better now | 11 | 3
  Much better now | 8 | 8

14. Secondary Outcome: Patient Global Assessment: Current Interfering Side Effects Versus Pain Relief During Previous Tramadol Treatment at Week 12
Description: Patients who have previously taken tramadol HCl were asked: "Compared to when you were previously taking tramadol, how have any side effects you have felt during this study interfered with your day-to-day activities?". Possible answers were: "Interfered much less now", "Interfered somewhat less now", "Same as before", "Interfered more now".
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Interfered much less now | 4 | 8
  Interfered somewhat less now | 2 | 1
  Same as before | 13 | 4
  Interfered more now | 3 | 0

15. Secondary Outcome: Physician Overall Rating: Overall Assessment at Week 12
Description: The physician was asked to indicate his overall assessment of the formulation the patient was taking using a 4-point Likert-scale dichotomized for the analysis: Very Effective, Effective, and Somewhat Effective were summarized to Effective; Ineffective remained unchanged.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Effective | 160 | 150
  Not effective | 1 | 3

16. Secondary Outcome: Physician Overall Rating: Effectiveness of Pain Control 24 Hours After the Most Recent Dose of Tramadol at Week 12
Description: The physician was asked to indicate the effectiveness of pain control 24 hours after the most recent dose of tramadol using a 4-point Likert-scale, dichotomized for the analysis: Very Effective, Effective, Somewhat Effective were summarized to Effective; Ineffective remained unchanged.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
participants
  Effective | 160 | 151
  Not effective | 1 | 2

17. Secondary Outcome: Patient Diary: Pain (Between Visit Means) at Week 12
Description: As part of the daily diary for the entire study, patients rated the arthritis pain in their worst knee using a five-point scale ranging from 1=none to 5=severe. Mean scores summarizing the entries of the preceding period were calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
Units on a scale | 2.74 (0.98) | 2.86 (1.08)

18. Secondary Outcome: Patient Diary: Stiffness (Between Visit Means) at Week 12
Description: As part of the daily diary for the entire study, patients rated the stiffness in their worst knee using a five-point scale ranging from 1=none to 5=severe. Mean scores summarizing the entries of the preceding period were calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
Units on a scale | 2.67 (0.96) | 2.82 (1.06)

19. Secondary Outcome: Patient Diary: Ability Getting Things Done (Between Visit Means) at Week 12
Description: As part of the daily diary for the entire study, patients rated their ability to get things done with their worst knee using a five-point scale ranging from: 1=No problem to 5=A lot of things didn't get done. Mean scores summarizing the entries of the preceding period were calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
Units on a scale | 2.41 (1.14) | 2.34 (1.18)

20. Secondary Outcome: Patient Diary: Difficulty With Walking (Between Visit Means) at Week 12
Description: As part of the daily diary for the entire study, patients rated their difficulty walking with their worst knee using a five-point scale ranging from 1=No problem to 5=Severe difficulty. Mean scores summarizing the entries of the preceding period were calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
Units on a scale | 2.79 (1.05) | 2.85 (1.11)

21. Secondary Outcome: Patient Diary: Difficulty With Stairs (Between Visit Means) at Week 12
Description: As part of the daily diary for the entire study, patients rated their difficulty with stairs with their worst knee using a five-point scale ranging from 1=No problem to 5=Severe difficulty. Mean scores summarizing the entries of the preceding period were calculated.
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Number analyzed (Participants) | 161 | 153
Units on a scale | 2.97 (1.14) | 3.10 (1.16)

ADVERSE EVENTS:
Arm/Group | Tramadol HCl Contramid® Once A Day | Tramadol HCl Twice a Day (SR)
Serious Adverse Events (participants affected / at risk) | 3/215 | 8/215
Other Adverse Events (participants affected / at risk) | 159/215 | 159/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol HCl Contramid® Once A Day (N=215) | Tramadol HCl Twice a Day (SR) (N=215)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Bladder Neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Disorder NOS (Nervous system disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Coronary Artery Insufficiency (Cardiac disorders) | 1 (1) | 0 (0)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Ischaemic Stroke NOS (Nervous system disorders) | 1 (1) | 0 (0)
Peritoneal Adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tramadol HCl Contramid® Once A Day (N=215) | Tramadol HCl Twice a Day (SR) (N=215)
Constipation (Gastrointestinal disorders) | 73 (136) | 65 (143)
Dizziness (Nervous system disorders) | 51 (85) | 65 (97)
Dry mouth (Gastrointestinal disorders) | 20 (28) | 10 (15)
Headache (Nervous system disorders) | 27 (37) | 38 (54)
Nausea (Gastrointestinal disorders) | 70 (121) | 73 (134)
Somnolence (Nervous system disorders) | 65 (113) | 46 (67)
Sweating increased (Skin and subcutaneous tissue disorders) | 16 (17) | 15 (25)
Vomiting (Gastrointestinal disorders) | 18 (24) | 31 (34)
Weakness (General disorders) | 24 (33) | 31 (47)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submitting results communications, the investigator shall allow Labopharm at least 30 days to review the proposed communication. If the proposed publication/disclosure risks Labopharm's ability to patent any invention related to the study, the publication or disclosure will be modified or delayed to allow Labopharm to seek patent protection. This statement does not give Labopharm any editorial rights other than to restrict the disclosure of Labopharm's confidential information